CLINICAL TRIAL: NCT04324723
Title: Behaviorally Enhanced Messages to Increase Medical Check-ups
Brief Title: Behaviorally Enhanced Messages to Increase Medical Check-ups(BEM-IMC)
Acronym: BEM-IMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kelly Ann Schmidtke (Other)
Collaborators: B4Development Foundation (Supreme Committee for Delivery and Legacy) (Unknown); Nudge Lebanon (Unknown); University of Warwick (Other)
Responsible Party: Sponsor-Investigator, Kelly Ann Schmidtke, Assistant Professor, University of Warwick
Organization: University of Warwick (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1
Record Dates: First submitted 2020-03-23; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: Health Seeking Behaviour; Opportunistic Screening; Randomised Controlled Trial
MeSH Terms: conditions — Hypertension; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researchers who called participants to ask if they sought further medical attention was not made aware of the participants' conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this group received a WhatsApp message reminding them to seek further medical attention for their measurement indicated hypertensive condition.
  Interventions: Behavioral: WhatsApp message
- Control (No Intervention): Participants in this group did not received a WhatsApp message reminding them to seek further medical attention for their measurement indicated hypertensive condition.

INTERVENTIONS:
Behavioral: WhatsApp message — The experimentally evaluated part of the intervention is a WhatsApp message.
  The message translated from Arabic to English appears below. "Dear [First name], Your BP reading during Beirut Marathon was [reading]. This indicates that you have elevated blood pressure. You should seek medical attention at your earliest convenience. Your wellbeing matters to us. Nudge Lebanon team"
  Arms: Intervention

SUMMARY:
The study had two stages. Stage 1 involved an opportunistic screening for hypertension conducted at the 2018 Beirut Marathon. During stage 1, participants whose measurements indicated hypertension were invited to take part in a RCT (randomized controlled trial). Stage 2 involved a RCT to evaluate the effectiveness of a behavioural intervention to increase the proportion of participants who sought further medical attention. The research team hypothesised that the intervention would increase the proportion of participants who sought further medical attention compared to a control group that did not receive the intervention.

This is a retrospective registration specifically focused on the RCT component of this study. The study was conducted by Nudge Lebanon in partnership with B4- development (formerly known as QBIU) and SmartScience. The RCT was not pre-registered because the collaborators were unaware that pre-registration would be necessary. The collaborators asked the University of Warwick to re-analyse and write the project up for publication after the study was complete. The University of Warwick is now seeking to retrospectively register the trial before submitting to an academic journal. The fact that this trial is retrospectively registered will be plainly stated in the manuscript and all analyses will be presented as exploratory.

DETAILED DESCRIPTION:
This study had two stages. Stage 1 involved an opportunistic screening and Stage 2 involved in RCT. This registration focuses on the RCT but both stages are described here.

Stage 1. The opportunistic screening for hypertension was conducted around the 2018 Beirut Marathon. Screening tents were set up at the marathon village during the four days leading up to the marathon (7-10 November), where runners collected necessary materials for the run and could take up the screening. An additional two tents were set up during the marathon day were spectators could take part. Participants indicated their consent for the screening before taking part. During their participation they completed surveys about their demographics and health information (including whether they were hypertensive). After they completed the survey, nurses and trained team members measured their blood pressure using calibrated equipment. Those participants whose measurements indicated hypertension were invited to participate in the RCT.

Stage 2. For the RCT participants were randomly assigned to either a intervention or control group in a 1:1 fashion. Participants in the intervention group were sent a WhatsApp message 25 days after the marathon reminding them to seek help for their hypertensive condition. Participants in the control group were not sent this message. Then one month later the researchers called all these participants to ask wither they sought further medical attention. The main outcome was whether participants self-reported seeking further medical attention.

The research objectives were as follows:

Stage 1 screening: Evaluate if the opportunistic screening increased people's awareness of their hypertensive condition.

Stage 2 RCT: Evaluate if the intervention increased the proportion of participants who sought further medical attention.

ELIGIBILITY:
Inclusion Criteria:

* objectively taken measurements at opportunistic screening indicated hypertension,
* provided informed consented to participate in the trial, and
* provided valid contact details for a smart phone with WhatsApp messenger

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Self-reported seeking of further medical attention. | Response taken 56 days after the opportunistic screening (1 = Yes-sought further medical attention, 0 = No)
  If participants tell the researcher that they sought further medical attention via a phone call they received approximately 1 month after the WhatsApp messages were sent to participants.

SECONDARY OUTCOMES:
Self-reported Hypertension | A survey response taken at the opportunistic screening.(1 = Yes-experiencing hypertension, 0 = No)
  Whether participant says in a pre-intervention survey that they are experiencing hypertension
Self-reported Diabetes | A survey response taken at the opportunistic screening.(1 = Yes-experiencing diabetes, 0 = No)
  Whether participant says in a pre-intervention survey that they are experiencing diabetes
Self-reported High Cholesterol | A survey response taken at the opportunistic screening.(1 = Yes-experiencing high cholesterol, 0 = No)
  Whether participant says in a pre-intervention survey that they are experiencing high cholesterol.
Systolic blood pressure (SBP) | An objective measure taken at the opportunistic screening using an Omron 5 Series BP742N blood pressure monitor
  Objectively measured at screening event
Diastolic blood pressure (DBP) | An objective measure taken at the opportunistic screening using an Omron 5 Series BP742N blood pressure monitor
  Objectively measured at screening event

OTHER OUTCOMES:
Heart rate | An objective measure taken at the opportunistic screening using an Omron 5 Series BP742N blood pressure monitor
  Objectively measured at screening event
year of birth | A survey response taken at the opportunistic screening.
  Year indicated in pre-intervention survey
Height in cm | A survey response taken at the opportunistic screening.
  Height indicated in pre-intervention survey
Weight in kg | A survey response taken at the opportunistic screening.
  Weight indicated in pre-intervention survey
Known family history of hypertension | A survey response taken at the opportunistic screening.
  Knowledge of family history indicated in pre-intervention survey
Know that high blood pressure could cause health problems | A survey response taken at the opportunistic screening.
  Knowledge of blood pressure health problems indicated in pre-intervention survey
knew that SBP measures over 140 mm Hg and DBP measures over 90mmHg (millimeters of mercury) were the diagnostic thresholds for stage II hypertension that may require treatment | A survey response taken at the opportunistic screening.
  Knowledge of diagnostic thresholds indicated in pre-intervention survey
Self-reported blood pressure checking | A survey response taken at the opportunistic screening. (1 = Yes-blood pressure checking, 0 = No)
  Self-reported blood pressure checking
Self-reported cholesterol checking | A survey response taken at the opportunistic screening. (1 = Yes-cholesterol checking, 0 = No)
  Self-reported cholesterol checking
Self-reported diabetes checking | A survey response taken at the opportunistic screening.(1 = Yes-diabetes checking, 0 = No)
  Self-reported diabetes checking
Self-reported attends regular physical check-ups | A survey response taken at the opportunistic screening.(1 = Yes-attends regular checkups, 0 = No)
  Self-reported attends regular physical check-ups
Self-reported uses alcohol | A survey response taken at the opportunistic screening.(1 = Yes-consumes alcohol, 0 = No)
  Self-reported uses alcohol
Self-reported smoking | A survey response taken at the opportunistic screening.(1 = Yes-smokes, 0 = No)
  Self-reported smoking

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Makki, PhD, Principal Investigator — B4Development Foundation
Locations (1):
- Nudge Lebanon. 3rd Floor, GS Building, Sit Nasab Street, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
The research team will cannot make identifiable individual participant data available.
  The de-identified participant data used in this papers analyses can be made available by contacting Kelly Ann Schmidtke (ORCID identifier: 0000-0001-5993-0358) and can be reused for further analyses.